CLINICAL TRIAL: NCT06592989
Title: A Clinical Study of Sorafenib Combined With Gefitinib for the Treatment of Pancreatic Neuroendocrine Tumor Patients Who Have Progressed After Previous Treatment
Brief Title: A Clinical Study of Sorafenib Combined With Gefitinib for the Treatment of pNET
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiuliang Yan, MD, Attending physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 20240625030921977
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Neuroendocrine Neoplasm; Sorafenib; Gefitinib
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Sorafenib; Gefitinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: This study is a single arm design, with only one experimental group set up. Medication plan and cycle: oral administration. Sorafenib: once a day, 250mg each time. Gefitinib: once a day, 250mg each time. Every 4 weeks is a treatment cycle.
  Interventions: Drug: sorafenib, gefitinib

INTERVENTIONS:
Drug: sorafenib, gefitinib — Sofantinib: 250mg, QD, oral; Gefitinib: 250mg, QD, oral.
  Other Names: No.

SUMMARY:
The incidence rate of pancreatic neuroendocrine neoplasms (pNENs) is increasing year by year. According to the statistical results of the SEER (Surveillance, Epidemiology, and End Results) database, the incidence rate of pNENs increased from 0.27/100000 to 1/100000 from 2000 to 2016, with a median overall survival time of 68 months. The 5-year overall survival rates of localized, locally advanced, and metastatic pNENs were 83%, 67%, and 28%, respectively. pNENs are gradually gaining attention and importance from the medical community. The existing therapeutic drugs for neuroendocrine tumors include somatostatin analogues, recombinant human interferon injections, chemotherapy drugs, and molecular targeted drugs.

Although these drugs can prolong patients' PFS to some extent, there is a common problem of low objective response rates. In recent years, sunitinib and everolimus have been approved for targeted therapy in patients with pancreatic neuroendocrine neoplasms , but their clinical efficacy is still limited. The study by Panzuto et al. showed that the median PFS for first-line treatment of advanced well differentiated pancreatic neuroendocrine neoplasms was 13.9 months, with an ORR of 14.9%. After imaging progression of the disease, the median PFS after second-line treatment was 15 months, and the ORR of only 5.5%. There is currently no effective treatment for patients with disease progression or drug resistance after undergoing existing treatment ways.

Therefore, there is a huge clinical demand for the treatment of pNEN patients worldwide, and effective drugs are urgently needed to benefit these patients.

Our previous research found that pathways in tumor were significantly affected in pNENs and liver metastases and EGFR tyrosine kinase inhibitor resistance and transcriptional dysregulation in tumor were unique to liver metastasis through KEGG pathway analysis; Meanwhile, GO Biological Processes analysis emphasizes those signaling pathways closely related to tyrosine phosphorylation, DNA repair, and cell cycle regulation, especially in liver metastases. Xiao et al. found that epidermal growth factor receptor (EGFR) was enriched in high glycosylation pNENs using RNA-seq. EGFR was expressed in 21.2% of pNENs using immunohistochemistry and associated with poor overall survival. Therefore, the study from Xiao et al. demonstrates that EGFR may be a potential therapeutic target for pNENs. This is consistent with our previous findings that the EGFR signaling pathway plays an important role in pNENs with liver metastases.

Due to the heterogeneity and complexity of tumors, the efficacy of monotherapy or blocking a single signaling pathway may be limited or this treatment method may easily develop drug resistance. The existing anti-tumor targeted drugs block tumor angiogenesis by inhibiting vascular endothelial growth factor (VEGF) and fibroblast growth factor (FGF). Colony-stimulating factor 1 receptor (CSF1R) is an important signaling pathway associated with the survival and function of tumor associated macrophages (TAMs). Inhibiting CSF1R can regulate the activity of macrophages, improve the immune microenvironment, promote immune response, and activate the body's immune function. Sofantinib is a novel oral tyrosine kinase inhibitor which exerts dual effects of anti-tumor angiogenesis and immune regulation by targeting VEGFR, FGFR1, and CSF1R, resulting in synergistic anti-tumor activity. In December 2020 and June 2021, sorafenib was approved in China as a monotherapy for unresectable locally advanced or metastatic, well differentiated extrapancreatic and pancreatic neuroendocrine neoplasms.

However, in a multicenter, single blind, open label, phase Ib/II clinical trial, the objective response rate for pNENs patients was only 19%. There is currently no effective treatment available for patients with disease progression or drug resistance after undergoing existing treatment regimens. Therefore, there is an urgent need to seek new treatment methods to improve the therapeutic effect of pNENs. Based on our previous research results and relevant literature reports, we speculate that the combination of sorafenib and EGFR inhibitor gefitinib may improve the therapeutic effect of pNENs patients.

DETAILED DESCRIPTION:
Neuroendocrine neoplasms (NENs) are heterogeneous tumors originating from peptidogenic neurons and neuroendocrine cells. Most commonly found in the digestive tract or lungs, it can be a benign or malignant tumor. According to their origin, neuroendocrine neoplasms are usually divided into pancreatic neuroendocrine neoplasms and non pancreatic neuroendocrine neoplasms. Approved targeted therapy drugs include sunitinib and everolimus, used to treat pancreatic neuroendocrine neoplasms or highly differentiated non functional gastrointestinal or pulmonary neuroendocrine neoplasms. The gastrointestinal tract and pancreas are home to 12 and 4 types of neuroendocrine cells, respectively, and are the most common sites of NEN occurrence, accounting for approximately 55% to 70% of all NENs. The incidence rate of neuroendocrine neoplasms from gastrointestinal tract and pancreas is about 5.25/100000, which is the second common tumor of gastrointestinal tract. In China, the ratio of incidence rate and prevalence of neuroendocrine neoplasms is estimated to be 4.4, lower than 7.4 in the United States.

In 2018, there were 19000 newly diagnosed cases of neuroendocrine neoplasms in the United States. It is noteworthy that compared with other tumors, the survival period of patients with neuroendocrine neoplasms is relatively long. Therefore, although the incidence rate of neuroendocrine neoplasms is relatively low, the patient population is relatively large. In addition, it is estimated that there were approximately 141000 neuroendocrine neoplasm patients in the United States in 2018, of which over 90%, or 132000 patients, were non pancreatic neuroendocrine neoplasm patients. In China, there were approximately 67600 newly diagnosed cases of neuroendocrine neoplasms in 2018. According to China's incidence to prevalence ratio, there may be as many as 300000 patients with neuroendocrine neoplasms in China. It is estimated that about 80% of patients with neuroendocrine neoplasms in China are non pancreatic neuroendocrine neoplasm patients. Octreotide and Lancreotide, which belong to Somatostatin Analogues SSAs, can alleviate symptoms such as flushing and diarrhea caused by carcinoid syndrome and have been widely used in clinical practice. In a phase III clinical study comparing long-acting octreotide LAR with placebo in the treatment of 85 cases of metastatic colorectal cancer NENs (PROMID), octreotide LAR significantly prolonged the time to disease progression (TTP) in patients: Octreotide LAR group at 14.3 months and placebo group at 6 months (p=0.000072). A systematic analysis report shows that after combination therapy with long-acting octreotide and other therapies (including everolimus, peptide receptor radionuclide therapy, bevacizumab, interferon, etc.), 85% of patients' diseases were controlled, with PFS ranging from 15 months to 16.4 months and OS ranging from 25 months to 61.9 months. SSAs are well tolerated drugs with few side effects, usually mild, and do not require discontinuation[5].

The incidence rate of pancreatic neuroendocrine neoplasms (pNENs) is increasing year by year. According to the statistical results of the Surveillance, Epidemiology, and End Results (SEER) database, the incidence rate of pNENs increased from 0.27/100000 to 1/100000 from 2000 to 2016, with a median overall survival time of 68 months, and the 5-year overall survival rates (OS) of localized, locally advanced, and metastatic pNENs were 83%, 67%, and 28% respectively. pNENs are gradually attracting attention and importance from the medical community. The existing therapeutic drugs for neuroendocrine neoplasms include growth hormone inhibitors, recombinant human interferon injections, chemotherapy drugs, and molecular targeted drugs. Although these drugs can to some extent prolong patients' PFS, there is a common problem of low objective response rates. In recent years, sunitinib and everolimus have been approved for targeted therapy in patients with pancreatic neuroendocrine tumors, but their clinical efficacy is still limited. The study from Panzuto et al. showed that the median PFS for first-line treatment of advanced well differentiated pancreatic neuroendocrine neoplasms was 13.9 months, with an ORR of 14.9%. When imaging progression occurred and second-line treatment was adopted, the median PFS after second-line treatment was 15 months, with an ORR of only 5.5%. There is currently no effective treatment for patients with disease progression or drug resistance after existing treatments.

Therefore, there is a huge clinical demand for the treatment of pancreatic neuroendocrine neoplasm patients both domestically and globally, and effective drugs are urgently needed to benefit the vast number of patients.

Our previous research found that tumor signaling pathways are significantly affected in pancreatic neuroendocrine neoplasms and liver metastasis through KEGG pathway analysis. EGFR tyrosine kinase inhibitor resistance and transcriptional dysregulation in tumors are unique to liver metastasis; Meanwhile, GO biological process analysis emphasizes signaling pathways closely related to tyrosine phosphorylation, DNA repair, and cell cycle regulation. Xiao et al. found that RNA seq was used to enrich epidermal growth factor receptor (EGFR) in high glycosylated pancreatic neuroendocrine neoplasms. Immunohistochemical staining revealed that 21.2% of pancreatic neuroendocrine tumors expressed EGFR, which was associated with low overall survival rate (P=0.020). Therefore, Xiao et al. believe that EGFR may be a potential therapeutic target for pancreatic neuroendocrine neoplasms. This is consistent with our previous findings that the EGFR signaling pathway plays an important role in pancreatic neuroendocrine neoplasms with liver metastasis.

Due to the heterogeneity and complexity of tumors, the efficacy of monotherapy or blocking a single signaling pathway may be limited. The existing targeted anti-tumor drugs block tumor angiogenesis by inhibiting vascular endothelial growth factor (VEGF) and fibroblast growth factor (FGF). Colony stimulating factor 1 receptor (CSF1R) is an important signaling pathway associated with the survival and function of tumor associated macrophages (TAMs). Inhibiting CSF1R can regulate the activity of macrophages , improve the immune microenvironment, promote immune response in the body, and activate immune function. Sofantinib is a novel oral tyrosine kinase inhibitor that exerts dual effects of anti angiogenesis and immune regulation by targeting vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR1), and colony-stimulating factor 1 receptor (CSF1R) kinases, resulting in synergistic anti-tumor activity. In December 2020 and June 2021, sorafenib was approved in China as a monotherapy for unresectable locally advanced or metastatic, well differentiated extrapancreatic and pancreatic neuroendocrine neoplasms. However, in a multicenter, single blind, open label, phase Ib/II clinical trial, the objective response rate for pancreatic neuroendocrine tumor patients was only 19%, and there is no effective treatment for patients with disease progression or drug resistance after existing treatment regimens. Therefore, there is an urgent need to seek new treatment methods to improve the therapeutic effect of pancreatic neuroendocrine neoplasms.

There is a study showing that dual inhibition of epidermal growth factor receptor and vascular endothelial growth factor pathways may delay therapeutic resistance in advanced non-small cell lung cancer (NSCLC). Bevacizumab plus erlotinib significantly improved PFS in patients with untreated metastatic EGFR-mutated NSCLC. Based on previous research results and relevant literature reports, we speculate that the combination of sorafenib and EGFR inhibitors gefitinib may improve the treatment efficacy of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a full understanding of this study and voluntarily sign an informed consent form;
2. Age ≥ 18 years old and age ≤ 80 years old;
3. Patients with pancreatic neuroendocrine tumors diagnosed by histopathology or cytology, who have progressed after previous treatments such as SSA, targeted therapy, and chemotherapy (all grades of pancreatic neuroendocrine tumors and neuroendocrine cancers are allowed to be included);
4. According to the criteria for evaluating the efficacy of solid tumors (RECIST V1.1), there should be at least one measurable lesion;
5. At least 7 days have passed since the end of the last systemic treatment, and palliative radiotherapy for localized areas is allowed. It has been completed for more than 4 weeks;
6. Expected survival time ≥ 12 weeks;
7. Researchers estimate that patients can benefit from it;
8. The patients have sufficient organ and bone marrow function;
9. Male or female patients with fertility voluntarily use effective contraceptive methods, such as double barrier contraception, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and within 6 months of the last study medication. All female patients will be considered to have fertility unless they have undergone natural menopause, artificial menopause, or sterilization surgery (such as hysterectomy, bilateral adnexectomy, or radiation ovarian irradiation).

Exclusion Criteria:

1. Other malignant tumors have been diagnosed in the past 5 years, except for effectively treated skin basal cell carcinoma, skin squamous cell carcinoma, or effectively resected cervical carcinoma in situ, breast cancer;
2. Simultaneously receiving other investigational drugs or approved or investigational anti-tumor treatments;
3. Patients with contraindications to experimental drugs (such as active bleeding, ulcers, intestinal perforation, intestinal obstruction, uncontrolled hypertension, III-IV grade heart failure, within 30 days after major surgery, severe liver and kidney dysfunction, etc.);
4. The patient currently has any diseases or conditions that affect drug absorption, or the patient is unable to take oral medication;
5. Confirmed allergy to any component of the investigational drug and/or its excipients;
6. Pregnant (positive pregnancy test before medication) or breastfeeding women;
7. Patients with large amounts of pleural effusion or ascites requiring drainage;
8. Any other disease with clinically significant metabolic abnormalities, physical examination abnormalities, or laboratory examination abnormalities. According to the researcher's judgment, it is suspected that the patient has a certain disease or condition that is not suitable for the use of the study drug (such as having seizures and requiring treatment), or that it will affect the interpretation of the study results, or put the patient in a high-risk situation;
9. Have taken medication containing components of Hypericum perforatum within 3 weeks prior to the first study medication. Or have taken other strong inducers or inhibitors of CYP3A4 within the previous 2 weeks;
10. According to the judgment of the investigator, the subject has other factors that may lead to the forced termination of this study or are not suitable for inclusion, such as other serious concomitant diseases (such as severe diabetes, thyroid disease, spinal cord compression, superior vena cava syndrome, mental illness), serious laboratory examination abnormalities, accompanied by family or social factors, which will affect the safety of the subject, or the collection of data and samples).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic neuroendocrine neoplasms diagnosed by histopathology or cytology show progression after previous treatments such as SSA, targeted therapy, chemotherapy, and so on.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate | Baseline examination, then every 8 weeks until 2 years
  Objective response rate refers to the proportion of patients whose tumor has shrunk to a certain extent and maintained it for a certain period of time, including cases of CR and PR. The RECIST 1.1 criteria are used to assess objective tumor response. The subjects must have measurable tumor lesions at baseline, and the efficacy evaluation criteria are divided into complete response (CR), partial response (PR), stable disease(SD), and progressive disease (PD) according to the RECIST 1.1 criteria.
progression free survival | Researchers conduct survival assessments every 12 weeks until 2 years.
  Progression free survival refers to the period from the date of treatment until the first occurrence of disease progression or death from any cause.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the combination therapy of sorafenib and gefitinib. | 2 years.
  According to NCICTCAE5.0, evaluate the number of participants with treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jiuliang Yan, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Jiang Long, M.D., Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Throughout the entire research period.
Access Criteria: Researchers studying pancreatic neuroendocrine tumors can apply to share relevant data. But the applicant's identification is required.

REFERENCES:
- [Result] Hofland J, Kaltsas G, de Herder WW. Advances in the Diagnosis and Management of Well-Differentiated Neuroendocrine Neoplasms. Endocr Rev. 2020 Apr 1;41(2):371-403. doi: 10.1210/endrev/bnz004. PMID 31555796
- [Result] Del Rivero J, Perez K, Kennedy EB, Mittra ES, Vijayvergia N, Arshad J, Basu S, Chauhan A, Dasari AN, Bellizzi AM, Gangi A, Grady E, Howe JR, Ivanidze J, Lewis M, Mailman J, Raj N, Soares HP, Soulen MC, White SB, Chan JA, Kunz PL, Singh S, Halfdanarson TR, Strosberg JR, Bergsland EK. Systemic Therapy for Tumor Control in Metastatic Well-Differentiated Gastroenteropancreatic Neuroendocrine Tumors: ASCO Guideline. J Clin Oncol. 2023 Nov 10;41(32):5049-5067. doi: 10.1200/JCO.23.01529. Epub 2023 Sep 29. PMID 37774329
- [Result] Yao JC, Fazio N, Singh S, Buzzoni R, Carnaghi C, Wolin E, Tomasek J, Raderer M, Lahner H, Voi M, Pacaud LB, Rouyrre N, Sachs C, Valle JW, Fave GD, Van Cutsem E, Tesselaar M, Shimada Y, Oh DY, Strosberg J, Kulke MH, Pavel ME; RAD001 in Advanced Neuroendocrine Tumours, Fourth Trial (RADIANT-4) Study Group. Everolimus for the treatment of advanced, non-functional neuroendocrine tumours of the lung or gastrointestinal tract (RADIANT-4): a randomised, placebo-controlled, phase 3 study. Lancet. 2016 Mar 5;387(10022):968-977. doi: 10.1016/S0140-6736(15)00817-X. Epub 2015 Dec 17. PMID 26703889
- [Result] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057
- [Result] Rinzivillo M, De Felice I, Magi L, Annibale B, Panzuto F. Octreotide long-acting release (LAR) in combination with other therapies for treatment of neuroendocrine neoplasia: a systematic review. J Gastrointest Oncol. 2021 Apr;12(2):845-855. doi: 10.21037/jgo-20-292. PMID 34012671
- [Result] Sonbol MB, Mazza GL, Mi L, Oliver T, Starr J, Gudmundsdottir H, Cleary SP, Hobday T, Halfdanarson TR. Survival and Incidence Patterns of Pancreatic Neuroendocrine Tumors Over the Last 2 Decades: A SEER Database Analysis. Oncologist. 2022 Jul 5;27(7):573-578. doi: 10.1093/oncolo/oyac049. PMID 35348774
- [Result] Panzuto F, Andrini E, Lamberti G, Pusceddu S, Rinzivillo M, Gelsomino F, Raimondi A, Bongiovanni A, Davi MV, Cives M, Brizzi MP, Persano I, Zatelli MC, Puliafito I, Tafuto S, Campana D. Sequencing Treatments in Patients with Advanced Well-Differentiated Pancreatic Neuroendocrine Tumor (pNET): Results from a Large Multicenter Italian Cohort. J Clin Med. 2024 Apr 3;13(7):2074. doi: 10.3390/jcm13072074. PMID 38610840
- [Result] Xu M, Yan J, Hu B, Wu C, Gu H, Qi Z, Chen T, Yang W, Zheng Y, Dong H, Sheng W, Long J. Evolutionary Trajectories of Primary and Metastatic Pancreatic Neuroendocrine Tumors Based on Genomic Variations. Genes (Basel). 2022 Sep 4;13(9):1588. doi: 10.3390/genes13091588. PMID 36140756
- [Result] Xiao Z, Xu H, Strosberg JR, Lu R, Zhu X, Deng S, Ding L, Ni Q, Warshaw AL, Yu X, Luo G. EGFR is a potential therapeutic target for highly glycosylated and aggressive pancreatic neuroendocrine neoplasms. Int J Cancer. 2023 Jul 1;153(1):164-172. doi: 10.1002/ijc.34499. Epub 2023 Mar 17. PMID 36891979
- [Result] Syed YY. Surufatinib: First Approval. Drugs. 2021 Apr;81(6):727-732. doi: 10.1007/s40265-021-01489-y. PMID 33788183
- [Result] Xu J, Li J, Bai C, Xu N, Zhou Z, Li Z, Zhou C, Jia R, Lu M, Cheng Y, Mao C, Wang W, Cheng K, Su C, Hua Y, Qi C, Li J, Wang W, Li K, Sun Q, Ren Y, Su W. Surufatinib in Advanced Well-Differentiated Neuroendocrine Tumors: A Multicenter, Single-Arm, Open-Label, Phase Ib/II Trial. Clin Cancer Res. 2019 Jun 15;25(12):3486-3494. doi: 10.1158/1078-0432.CCR-18-2994. Epub 2019 Mar 4. PMID 30833272
- [Result] Zhou Q, Xu CR, Cheng Y, Liu YP, Chen GY, Cui JW, Yang N, Song Y, Li XL, Lu S, Zhou JY, Ma ZY, Yu SY, Huang C, Shu YQ, Wang Z, Yang JJ, Tu HY, Zhong WZ, Wu YL. Bevacizumab plus erlotinib in Chinese patients with untreated, EGFR-mutated, advanced NSCLC (ARTEMIS-CTONG1509): A multicenter phase 3 study. Cancer Cell. 2021 Sep 13;39(9):1279-1291.e3. doi: 10.1016/j.ccell.2021.07.005. Epub 2021 Aug 12. PMID 34388377